CLINICAL TRIAL: NCT00373542
Title: A 12-Week, Multi-Center, Double-Blind, Placebo-Controlled, Parallel Group, Flexible Dose Polysomnography Study of Ropinirole Controlled Release for Restless Legs Syndrome (RLS) in RLS Patients With Sleep Disturbance and Periodic Limb Movements (PLM) During Sleep
Brief Title: 12-week Polysomnography Study of Ropinirole Controlled Release for Restless Legs Syndrome
Acronym: (CR-RLS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRL103660
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Restless Legs Syndrome (RLS); Restless Legs Syndrome
Keywords: Restless Legs Syndrome; ropinirole; polysomnography; RLS; PSG
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ropinirole CR-RLS

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ropinirole CR-RLS in the treatment of patients with Restless Legs Syndrome and associated sleep disturbance and period limb movements during sleep.

ELIGIBILITY:
Inclusion criteria:

* provided written informed consent.
* Diagnosed with primary RLS using the International RLS Study Group Diagnostic Criteria with a total score of 20 or greater on the International RLS (IRLS) Rating Scale and significant sleep disturbance indicated on Item 4 of the IRLS rating scale.
* Have evening and nighttime symptoms of RLS, significant sleep impairment due to RLS symptoms, and symptoms requiring treatment prior to bedtime, but no earlier than 5:00PM.
* Sleep efficiency <85% OR Latency to persistent sleep >20 minutes.

Exclusion criteria:

* Secondary RLS
* Primary sleep disorder
* Have any medical conditions that may impact efficacy assessments or that may present a safety concern.
* Pregnant or lactating or women of child-bearing potential who are not practicing an acceptable method of birth control.
* Use of any prohibited medication.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Periodic Limb Movements in Sleep associated with Arousal/hour of sleep (PLMAI) at Week 12 Change from baseline in sleep Latency at Week 12. | 12 Weeks

SECONDARY OUTCOMES:
Assess safety, tolerability, polysomnography efficacy measures, and patient reported outcomes. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- United States (44):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Greenwood, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Danville, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Brighton, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Lafayette Hill, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Walla Walla, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: RRL103660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: RRL103660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: RRL103660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: RRL103660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: RRL103660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: RRL103660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: RRL103660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register